CLINICAL TRIAL: NCT06824207
Title: Repeated Cross Sectional Surveillance Study To Determine the Respiratory Syncytial Virus (RSV) Immunization Rates in German Infants During Three RSV Seasons
Brief Title: Repeated Cross Sectional Surveillance Study To Determine the Respiratory Syncytial Virus (RSV) Immunization Rates in German Infants
Acronym: Vakzimeter RSV
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: RSV00093
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Syncytial Virus Immunization
Keywords: RSV; RSV Immunization Rates; Nirsevimab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Catch-Up Cohort: Parents of infants born between April and September
- In-Season Cohort: Parents of infants born between October and March

SUMMARY:
In June 2024, the German Standing Committee on Vaccination (STIKO) recommended the universal immunization of infants with nirsevimab during their first RSV season. Nirsevimab is a long-acting monoclonal antibody designed to provide passive immunity against RSV, significantly reducing the risk of severe RSV disease in infants. This recommendation marks the 2024/25 season as the first in which nirsevimab is broadly implemented for all infants in Germany.

Despite the introduction of this new prevention measure, there is currently no timely monitoring system for immunization rates. Understanding the uptake and coverage of nirsevimab is crucial for evaluating its impact on public health and guiding future vaccination strategies. Therefore, this study aims to monitor the national immunization rates of nirsevimab in children under one year of age during the initial seasons of its widespread use.

The primary objective of this study is to determine the Nirsevimab immunization rate in eligible infants in their first RSV-season in Germany. The study will focus on:

1. Assessing the immunization rates among eligible infants (according to STIKO recommendation) in their first RSV-season in Germany (i.e. across all geographies)
2. Assessing the immunisation rates among the "catch-up cohort", i.e. all infants born between April and September. For these infants, the STIKO recommends immunization with nirsevimab in early autumn.
3. Assessing the immunization rate among the "in-season cohort", i.e. all infants born during the RSV season between October and March. For these newborns, the STIKO recommends immunization with Nirsevimab shortly after birth, preferably during the second "well-baby visit" at the age of 3-10 days of life.

ELIGIBILITY:
Inclusion Criteria:

* Be a parent of an infant born between April 2024/25/26 and March 2025/26/27, respectively
* Reside in Germany at the time of survey completion
* Be at least 18 years old at the time of survey completion.
* Agree with privacy policy and AE (Adverse Event) reporting requirements before proceeding with the survey.
* Read and agree to the ICF (Informed Consent Form) by ticking a box before proceeding with the survey.

Exclusion Criteria:

* Participation in the study (= completed the survey) in a previous wave of the current season.

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is conducted using various recruitment approaches, including but not limited to mailings, online panels, telephone contact, in person contact. The data i.e. respondents answers will be captured via an online questionnaire. The interviews will be conducted applying various methodologies e.g. self-completion (CAWI), assisted in person completion (F2F interviews), assisted telephone completion (CATI).
  The study will target a sample of parents of infants either born between April and September (catch-up cohort) or between October and March (in-season cohort). The study targets a representative distribution with regards to both aforementioned subgroups and regions.
  To achieve the primary objective in the representative sample of the German population of eligible parents, a needed sample size of approximately 2,400 participants in total per season is assessed. These are spread over a total of three waves per season, resulting in a sample size of 800 respondents per wave.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the nirsevimab immunization rates among eligible infants in both cohorts | Throughout Study (Approximatley 4 months)
  Descriptive analysis of nirsevimab immunization status (yes/no) will be performed using summary statistics, i.e., proportion of immunized infants among all enrolled infants per wave.

SECONDARY OUTCOMES:
Assessing the seasonal evolution of the nirsevimab immunization coverage rates among the two cohorts | Throughout Study (Approximatley 4 months)
  Descriptive analysis of nirsevimab immunization status over time will be performed using summary statistics, i.e., proportion of immunized infants among all enrolled infants per wave.
Assessing reasons for/against nirsevimab immunization | Throughout Study (Approximately 4 months)
  The analysis for any potential influencing factors will be based on descriptive analytics and complemented with bi-variate analytics where applicable
Assessing the nirsevimab immunization rates among subgroups | Throughout Study (Approximately 4 months)
  A descriptive analysis of immunization rates will be performed on subgroups such as: risk group (defined chronic condition or pre-term birth status), federal states and health insurance/Kassenärztliche Vereinigung, physician's association regions
Assessing the reliability of a demographic study | Throughout the Study (Approximately 4 months)
  Assessing reliability based on randomly sampled parent population using Computer-Assisted Web Interview (CAWI)/ Computer-Assisted Telephone Interview (CATI)/ face-to-face interviews for estimating immunization rates in Germany

CONTACTS AND LOCATIONS:
Locations (1):
- Germany, Germany, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org